CLINICAL TRIAL: NCT03726801
Title: Prevention of Body Image Disorder by Nurse Intervention on the Patient and Family Prior to Breast and Colon Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Natalia Mudarra García, principal investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NATALIA MUDARRA GARCÍA
Record Dates: First submitted 2018-09-25; First posted 2018-11-01 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Body Image Disorder
Keywords: Body image; Conservative surgery; Quality of life; Breast cancer; Mastectomy; Ostomy; Colon cancer; Self esteem
MeSH Terms: conditions — Body Dysmorphic Disorders; Breast Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a non-blinded, randomized, controlled clinical trial consisting of 64 participants, which aims to assess the effectiveness of a nursing intervention for family members and patients prior to surgery to prevent body image disorder in breast cancer operated subjects. or colon (32 participants), compared to the intervention limited only to patients (32 participants).
Who Masked: Investigator
Masking Description: This is a non-blinded, randomized, controlled clinical trial consisting of 64 participants, which aims to assess the effectiveness of a nursing intervention for family members and patients prior to surgery to prevent body image disorder in breast cancer operated subjects. or colon (32 participants), compared to the intervention limited only to patients (32 participants).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stratum C (Experimental): N 32 C
  Women who are going to be mastectomized, conservate surgery and ostomy who attend the health education together with their immediate family member prior to surgery
  Interventions: Other: HEALTH EDUCATION
- Stratum E (Placebo Comparator): N 32 E
  Patients who are going to be subjected to a mastectomized, conservate surgery and ostomy who come alone to the health education prior to surgery
  Interventions: Other: HEALTH EDUCATION

INTERVENTIONS:
Other: HEALTH EDUCATION — The nursing intervention prior to surgery: (breast and colon cancer):
  1. First phase: At first these subjects suffered a great emotional impact after knowing the diagnosis, which could generate intense anxiety reactions.
  2. Second phase or phase of coping, in which they begin to be aware of their illness and the future changes they will suffer in their body. In this phase they react with fear, anger, anger, denial, ...
  3. Third phase or phase of adaptation to the new situation, where there is a decrease in previous emotional reactions, the patient being able to start up the resources learned to reduce their psychological discomfort.

SUMMARY:
This is a non-blinded, randomized, controlled clinical trial consisting of 64 participants, which aims to assess the effectiveness of a nursing intervention for family members and patients prior to surgery to prevent body image disorder in breast cancer operated subjects. or colon (32 participants), compared to the intervention limited only to patients (32 participants).

DETAILED DESCRIPTION:
Cancer is one of the most important public health problems on a global scale in the 21st century. The National Institute of Neoplastic Diseases highlights, among the most frequent neoplasms, prostate cancer, colon-rectum, lung in men and breast, colon-rectum in women.

One of the main treatments to be able to approach this type of tumors, such as breast and colorectal, is surgery. There are different surgical procedures (conservative surgery, mastectomy, ostomy) that, in a forceful way, affect the body image of the individual, sometimes generating extreme and painful situations. They are procedures that carry biopsychosocial implications and that generate a change in lifestyle.

A better psychological preparation and an effective health education of the patient prior to surgery (consisting of providing the information of the intervention, providing psychological support during the entire surgical process and reporting on the changes that will occur), balance the characteristic stressful trait of surgery, thus decreasing the level of anxiety of the individual.

In order for the patient to overcome this change in his body image, the role played by his immediate family member is fundamental, not only because it helps him improve the quality of life that he will have during the course of his illness, but also because an adequate emotional state can improve the patient's therapeutic response.

The objective of this study was to evaluate the body image disorder suffered by patients with breast and colorectal cancer after undergoing surgery, comparing the group that received a previous nursing intervention with their immediate family member, compared to the patients who received this intervention without him.

A randomized, non-blinded, controlled clinical trial was conducted. The study consisted of performing a nursing intervention prior to breast and colon surgery to both groups, giving health education divided into four phases: providing information on the disease, showing surgeries and similar experiences, explaining coping methods and reporting on techniques of relaxing.

ELIGIBILITY:
MOM:

Inclusion criteria:

* - Women over 18 years old.
* Oncological patients diagnosed with breast cancer (ductal carcinoma in situ, infiltrating ductal carcinoma, infiltrating lobular carcinoma, multicentric carcinoma, paget tumor ...), which are going to be subjected to surgery (mastectomy, lymphadenectomy, sentinel lymph node biopsy, surgery conservative ...).
* Not having received chemotherapy before surgery.
* Live with a direct family member.
* Not having received radiotherapy before surgery.
* Receive or not neoadjuvant hormone therapy.

Exclusion criteria:

* - Mens.
* Rejection of the surgical intervention.
* Non-cancer patient that will be operated on.
* Performing surgery in another hospital.
* Cancer patient diagnosed with breast cancer without surgical intervention.
* Refusal of the patient to know his diagnosis or impossibility to give his consent.
* Be submitted to tumor biopsy, without surgical intervention.

COLON:

* Inclusion criteria:

  * Women and men over 18 years of age.
  * Oncological patients diagnosed with colorectal cancer (adenocarcinoma of the lower rectum, adenocarcinoma of the middle rectum, colloid or mucinous adenocarcinoma), who are going to undergo surgery (colostomy, ileostomy ...).
  * Receive chemotherapy before or after surgery.
  * Receive radiotherapy before or after surgery.
  * Live with a direct family member.
* Exclusion criteria:

  * Rejection of surgical intervention.
  * Non-cancer patient that will be operated on.
  * Performing surgery in another hospital.
  * Oncological patient diagnosed with colon cancer without surgical intervention.
  * Refusal of patients to know their diagnosis or inability to give their consent.
  * Be submitted to tumor biopsy, without surgical intervention.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Average result in patients who have a body image disorder accompanied with or without a direct family member evaluated by the BIS Scale. | 16 months
  he alteration of the body image will be evaluated with the BIS SCALE after surgery, in the control group (patients who attend the nursing intervention prior to the same without family), and in the study group (patients who attend this intervention together with a direct family member). The Bis Scale has a score of 0 to 30 with 0 being no alteration of the body image and 30 a severe alteration.

SECONDARY OUTCOMES:
Average body image in all patients, to check the alterations that refer to perform a nursing intervention prior to surgery. | 16 months
  Alterations of the body image with the BIS Scale are measured in all patients to check if these alterations are reduced when performing an intervention prior to surgery. The Bis Scale has a score of 0 to 30 with 0 being no alteration of the body image and 30 a severe alteration.
Percentage of the self-esteem of the patients, differentiating whether or not they go with a direct family member, evaluated by the Rosenberg Scale. | 16 months
  Percentage of patients who have high self-esteem, average self-esteem and low self-esteem, differentiating whether they go with a direct relative or without him to the nursing intervention prior to surgery. This measurement is made to check if the family influences the patient's self-esteem. The Rosenberg scale has a score of 10 to 40 points: 30-40 high self-esteem, 26-29 average self-esteem and less than 25 low self-esteem.
Percentage of the Rosenberg scale in all patients, to check the self-esteem that patients refer to when performing a nursing intervention prior to surgery. | 16 months
  The percentages of self-esteem with the Rosenberg Scale are measured in all patients to see if self-esteem improves when performing a nursing intervention prior to surgery. The Rosenberg scale has a score of 10 to 40 points: 30-40 high self-esteem, 26-29 average self-esteem and less than 25 low self-esteem.
Average of the quality of life that patients have, differentiating whether or not they go with a direct family member, evaluated by the QLQBR23 Scale | 16 months
  The average of the QLQ Scale is calculated. BR23 - quality of life (concern for the future, sex practice, enjoyment of sex, breast symptoms, arm symptoms), differentiating whether patients with direct family members or without them go to the nursing intervention prior to surgery. This measurement is made to check if the family influences their quality of life. The QLQ BR 23 Scale have a score of 0 to 100 points, with a lower score being better functionality for worry about the future, symptoms of the breast and arm symptoms, and a lower score for worse functionality in sex enjoyment and sex practice.
Percentages of the Rosenberg Scale and average of the Bis Scale in all patients, to check whether the body image is related to self-esteem. | 16 months
  The percentages of the Rosenberg Scale and the means obtained with the BIS Scale are calculated. The relationship between these two scores obtained is checked to see if having greater alterations in body image is related to having low self-esteem. The Rosenberg scale has a score of 10 to 40 points: 30-40 high self-esteem, 26-29 average self-esteem and less than 25 low self-esteem. The Bis Scale has a score of 0 to 30 with 0 being no alteration of the body image and 30 a severe alteration.
Percentages in the Bis Scale and in the QLQ BR23 scale in all patients, to check if the body image is related to the quality of life. | 16 months
  The percentages of the Bis Scale and the QLQ BR23 Scale are calculated. The relationship between the two scores obtained is verified, to check if having greater alterations in body image is related to having quality of life. The Bis Scale has a score of 0 to 30 with 0 being no alteration of the body image and 30 a severe alteration.The QLQ BR 23 Scale have a score of 0 to 100 points, with a lower score being better functionality for worry about the future, symptoms of the breast and arm symptoms, and a lower score for worse functionality in sex enjoyment and sex practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Natalia Mudarra Garcia, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Criteria and Procedures for Breast Conserving Surgery. — https://www.google.com/search?safe=active&hl=es_419&source=hp&ei=1KfDW5r-J4WusAGWnqGgAQ&q=Fajdic+J%2C+Djurovic+D%2C+Gotovac+N%2C+Hrgovic+Z.+Criteria+and+Procedures+for+Breast+Conserving+Surgery.+Acta+Inform+Medica.+marzo+de+2013%3B21%281%29%3A16-9.+&oq=Fajdic+J%2C+Djurovic+D%2C+Gotovac+N%2C+Hrgovic+Z.+Criteria+and+Procedures+for+Breast+Conserving+Surgery.+Acta+Inform+Medica.+marzo+de+2013%3B21%281%29%3A16-9.+&gs_l=psy-ab.3...1459.1459.0.1980.3.2.0.0.0.0.0.0..1.0....0...1c.2.64.psy-ab..2.0.0.0...212.Mczz0xKChfk
- See also: Breast-conserving surgery versus modified radical mastectomy in treatment of early stage breast cancer: A retrospective study of 107 cases. — https://www.ncbi.nlm.nih.gov/pubmed/26323920
- See also: [Influence of the social context on the body image perception of women undergoing breast cancer surgery]. — https://www.ncbi.nlm.nih.gov/pubmed/24160199
- See also: Imagen corporal y autoestima en mujeres con cáncer de mama participantes en un programa de intervención psicosocial. — http://scielo.isciii.es/scielo.php?script=sci_arttext&pid=S1130-52742007000200002
- See also: Quality-of-life outcomes between mastectomy alone and breast reconstruction: comparison of patient-reported BREAST-Q and other health-related quality-of-life measures. — https://www.ncbi.nlm.nih.gov/pubmed/23897347
- See also: Percepción de la imagen corporal de la mujer intervenida de cáncer de mama y residente en la ciudad de Granada. — http://scielo.isciii.es/scielo.php?script=sci_abstract&pid=S0212-16112013000500012
- See also: The relationship between body image disturbance and distress in colorectal cancer patients with and without stomas. — https://www.ncbi.nlm.nih.gov/pubmed/21511069

DOCUMENTS (3):
  • Study Protocol (2018-09-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT03726801/Prot_001.pdf
  • Statistical Analysis Plan (2018-09-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT03726801/SAP_002.pdf
  • Informed Consent Form (2018-09-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT03726801/ICF_003.pdf